CLINICAL TRIAL: NCT02676440
Title: A Study to Measure the Effect of a Toothpaste Containing Zinc Citrate Trihydrate Used in Combination With a Serum Containing Zinc Sulphate Heptahydrate and a Standard Fluoride Toothpaste on Gingival Health Over a Six Month Period.
Brief Title: Effect of a Toothpaste and Serum Compared to Standard Fluoride Toothpaste on Gingival Health Over a Six Month Period.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: University of Bristol Dental Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ORL-GUM-2101
Record Dates: First submitted 2015-12-03; First posted 2016-02-08 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Healthy
Keywords: Oral Health
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Other): Toothpaste containing 1.11% Fluoride as Sodium Monofluorophosphate and Zinc Citrate Trihydrate Serum containing 0.17% Fluoride as Sodium Monofluorophosphate and Zinc Sulphate Heptahydrate
  Interventions: Other: Treatment
- Comparator (Other): Silica toothpaste 1350ppm F as Sodium Fluoride
  Interventions: Other: Comparator

INTERVENTIONS:
Other: Treatment — F13/T38
  Arms: Treatment
Other: Comparator — M26
  Arms: Comparator

SUMMARY:
This study is a double-blind, randomised, parallel group efficacy study. Up to 240 healthy female and male participants aged over 18 years will participate. There will be two groups of up to 120 participants. Participants will be randomised to the test groups according the allocation table prepared by the Statistician.

Participants will be enrolled on to the study according to the inclusion/exclusion criteria. After enrollment participants will have their teeth that have been allocated for assessment cleaned using a professional prophylaxis polish by the study dentist. The participants will then be provided with a standard cosmetic silica Fluoride toothpaste and a toothbrush to use at home, twice a day for up to four weeks. After this time they will return to the test site and have the baseline dental assessments. Participants will then be randomly allocated to one of the two test products which they will use at home, twice a day for the duration of the study. Dental assessments will be conducted after 13 and 26 weeks of product use at the study site.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18 years and over, of either gender and in good health.
* Be willing and physically able to carry out all study procedures.
* Be willing and competent (verbally and cognitively) to give written informed consent and complete a medical history form.
* Have at least 20 natural teeth including 5 teeth (excluding 3rd molars) in each quadrant
* Have at least 6 natural teeth assessable teeth in the Upper 4 to 4 region.
* Have a mean Modified Gingival Index (MGI) score of 2 at screening in the Upper 4 to 4 region.
* Not have had a scale and prophylaxis in the month prior to enrolment or have one scheduled prior to the end of the study.
* Be willing to use the test products for 6 months

Exclusion Criteria:

* Current participation in any other cosmetic trials, any dental clinical trials or clinical trials.
* Pregnant or nursing women.
* Medical condition and/or regular use of any medication which might affect the outcome of the study, as determined by the study dentist, principally a course of anti-inflammatory, antimicrobial or statin drugs
* Obvious signs of untreated caries or significant periodontal disease, which in the opinion of the Study Dentist, will affect either the scientific validity of the study or if the participants was to participate in the study would affect their wellbeing.
* Any participant who, in the judgement of the investigator, should not participate in the study.
* Full or partial dentures wearers.
* Current orthodontic treatment.
* Have oral piercings.
* Smokers or those who have a recent smoking history.
* Taking dietary supplements (e.g. multivitamins; antioxidants; fish oils).
* Any subject with a single MGI score of 4 in the any area of the mouth at any time point will be excluded.
* A subject will be excluded from the study if they have a MGI mouth mean of >2.75 at screening
* Any subject with a single MGI score of 3 at Baseline
* Use of non study oral care products, e.g. dental floss, chewing gum, mouth rinses during the pre treatment and test phases of the study.
* The subject is an employee of Unilever or a member of the study team.
* Taking a course of antimicrobial or anti-inflammatory drugs within 4 weeks of screening
* Those taking anti-histamine or anti-inflammatory medication in the 24 hours prior to the dental assessments
* Diabetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2015-07-03 (Actual); Primary Completion 2015-12-14 (Actual); Study Completion 2016-03-14 (Actual)

PRIMARY OUTCOMES:
Change in gingival condition as assessed using the Modified Lobene Gingival Index | 13 weeks
Change in gingival condition as assessed using the Saxton and van der Ouderaa bleeding index | 13 weeks
Change in gingival condition as assessed using the Modified Quigley and Hein plaque index | 13 weeks

SECONDARY OUTCOMES:
Change in gingival condition as assessed using the Modified Lobene Gingival Index | 26 weeks
Change in gingival condition as assessed using the Saxton and van der Ouderaa bleeding index | 26 weeks
Change in gingival condition as assessed using the Modified Quigley and Hein plaque index | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicola X West, BDS, Principal Investigator — Bristol Dental Hospital and School
Locations (1):
- Bristol Dental Hospital and School, Bristol, United Kingdom